CLINICAL TRIAL: NCT01896934
Title: Frontal Hypoperfusion Effects on Antidepressant Outcomes in Late-Life Depression (R21)
Brief Title: Frontal Hypoperfusion Effects on Antidepressant Outcomes in Late-Life Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Warren Taylor, Associate Professor of Psychiatry, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 130360; R21MH099218-01A1 (NIH)
Record Dates: First submitted 2013-07-01; First posted 2013-07-11 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2017-07-21 (Actual); Status verified 2017-06

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Antidepressants; Elderly; Geriatrics
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sertraline (Experimental): 50-200mg daily
  Interventions: Drug: Sertraline

INTERVENTIONS:
Drug: Sertraline — 50-200mg daily
  Other Names: Zoloft

SUMMARY:
The long-term goal of this line of research is to determine if decreased vascular reactivity and frontal hypoperfusion is associated with poor response antidepressants. Such perfusion deficits could contribute to antidepressant nonresponse as they would hinder improvements in dorsal system metabolism seen with antidepressant treatment. The objective of the current proposal is to determine if decreased vascular reactivity and frontal hypoperfusion in depressed elders predicts and persists with antidepressant nonremission. The investigators will pursue the primary aim testing the hypothesis that decreased reactivity and hypoperfusion, specifically in the dorsolateral prefrontal cortex and dorsal anterior cingulate cortex, predict antidepressant nonremission. The investigators will enroll 40 depressed elders who will complete clinical, cognitive, and MRI assessments before and after a 12-week open-label antidepressant trial of sertraline.

DETAILED DESCRIPTION:
The long-term goal of this line of research is to determine if in late-life depression (LLD), cerebrovascular dysregulation is predictive of antidepressant outcomes. The investigators hypothesize that vascular pathology resulting in reduced cerebrovascular reactivity contributes to frontocingulate hypoperfusion. Such pathology would impair neurovascular coupling and reduce the ability of the vasculature to improve frontocingulate perfusion during antidepressant treatment. Thus decreased cerebrovascular reactivity and perfusion may be a biomarker of antidepressant nonresponse. As an initial step in this research, the current study will utilize MRI arterial spin labeling (ASL) to examine if cerebrovascular reactivity deficits and resting cerebral blood flow (CBF) deficits predict antidepressant nonremission in LLD. The rationale for this proposal is that it will identify mechanisms by which vascular pathology may contribute to LLD. If the study hypotheses are correct, this crucial next step will support studies examining antidepressant properties of cardiovascular drugs that may reverse vascular pathology and improve perfusion.

The investigators will pursue our initial goal by examining ASL predictors of nonremission to a 12-week trial of sertraline. Forty LLD subjects will complete MRI, cognitive testing, and hyperintensity assessment. ASL measured CBF will be obtained during a hypercapnia challenge and at rest with room air. This will help determine if deficits in cerebrovascular reactivity (CVR) and/or resting and on-demand CBF measures predict nonremission.

AIM: To test for differences in CVR and CBF in dorsal frontal cognitive control regions between individuals who do and do not remit to a 12-week course of sertraline (defined as MADRS ≤ 7).

Hypothesis 1: Compared with remitters, during a hypercapnia challenge nonremitters will exhibit less CVR in the dlPFC and dAC.

Hypothesis 2: Compared with remitters, while breathing room air nonremitters will exhibit lower resting CBF in the dorsal anterior cingulate (dAC) and dorsolateral prefrontal cortex (dlPFC).

Exploratory Aim: To examine the relationship between ASL measures (CVR to hypercapnia and resting CBF during normoxia) and performance in cognitive domains implicated in LLD treatment outcomes. For this Aim, we will focus on functions involving the dlPFC and dAC, specifically executive function and processing speed.

The study will enroll patients from clinical referrals and response to advertisements. In these cases, potential participants will call our study contact number. Study staff will describe the study to them, including a description of the study entry criteria. Those who continue to be interested will then be scheduled for an evaluation. After scheduling, a study physician will review their electronic medical record to assure that potential subjects meet entry criteria.

Following policies of the Vanderbilt University Health System Institutional Review Board, written informed consent will be obtained and documented by the study's Research Coordinator before any study-related procedures are performed. The study coordinator will review study procedures and the consent form with each potential participant. Each individual may take as much time as they like to decide if they do or do not wish to participate. There is no randomization. All participants receive open-label sertraline.

An initial evaluation will determine eligibility, depression severity, and evaluate medical and psychiatric history. Participants will also complete a detailed battery assessing cognitive function. During this time they will also complete the one-hour MRI session, which includes measurement of cerebral perfusion and vascular reactivity.

They will then begin the 12-week trial of open-label sertraline, allowing titration up to the maximum dose of 200mg daily. At the end of the study participants will be referred for ongoing clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60 years or older.
2. Current diagnosis of major depressive disorder (DSM-IV-TR), single episode, recurrent or chronic, without psychotic features, as detected by MINI and clinical exam.
3. Minimum MADRS score ≥ 15.
4. Mini-Mental State Exam ≥ 22.
5. Ability to read and write English.

Exclusion Criteria:

1. Current or past diagnoses of other Axis I psychiatric disorders, including panic disorder and substance dependence.
2. Any use of illicit substances (such as marijuana or cocaine) or abuse of prescription medications (such as benzodiazepines or opiates) within the last three months.
3. Presence of acute suicidality
4. Current or past psychosis
5. Known primary neurological disorder, including dementia, brain tumors, epilepsy, Parkinson's disease, or demyelinating diseases
6. Chronic untreated medical disorders (including but not limited to hypertension, hyperlipidemia, fibromyalgia, hypothyroidism, or any other disorder) where treatment is warranted
7. Need for continuous oxygen use or any medical disorder where the hypercapnia challenge would be contraindicated or put the subject at increased risk. This would include active respiratory disease, chronic angina or other unstable cardiac conditions.
8. Any physical or intellectual disability affecting completion of assessments
9. MRI contraindications
10. Electroconvulsive therapy in last 6 months
11. Use of fluoxetine in the last 6 weeks. Occasional use of benzodiazepines or non-benzodiazepine sedatives (such as zolpidem, eszopiclone, or zaleplon) during the last month is allowable.
12. Known allergy or hypersensitivity to sertraline
13. A failed therapeutic trial of sertraline in the current depressive episode (defined as at least 6 weeks of treatment at a daily dose of 100mg or higher)
14. Current or planned psychotherapy

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2013-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Warren D Taylor, MD, MHSc, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants taking ineffective antidepressant medications underwent a washout period. 10 recruited individuals were withdrawn after screening for a) concomitant medications (N=2), b) depression not severe (N=4), c) MRI contraindications (N=4)
Period: Overall Study
Arm/Group | Sertraline
Started | 21
Completed | 19
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sertraline
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.05 (7.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 21
Montgomery-Asberg Depression Rating Scale [Mean (Standard Deviation); unit: units on a scale] — Depression rating scale, clinician rated, range 0-60, where higher scores indicate more severe depression
  units on a scale | 27.43 (4.80)
Quick Inventory of Depressive Symptoms [Mean (Standard Deviation); unit: units on a scale] — Depression rating scale, self-report, Range 0-27, where higher scores indicate more severe depression Population: Baseline data missing for 4 individuals (3 subject did not complete, 1 deviation where questionnaire was not provided to subject)
  units on a scale
    number analyzed (Participants) | 17
    (all) | 11.94 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Remission of Depression
Description: Montgomery-Asberg Depression Rating Scale (MADRS) is a measure of depression severity. This will be used to define remission as a score of 7 or less.
Time Frame: Week 12
Population: Individuals achieving remission of depression, defined as MADRS score of 7 or less.
Measure: Count of Participants; unit: Participants
Arm/Group | Sertraline
Number analyzed (Participants) | 21
Participants | 10

2. Secondary Outcome: Change in Clinician-rated Depression Severity
Description: Change in depression severity will be measured by the clinician-rated Montgomery Asberg Depression Rating Scale (MADRS), range of 0-60, with higher scores indicating more severe depression
Time Frame: Assessed every 2 weeks from baseline to week 12, change from baseline to week 12 is reported
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sertraline
Number analyzed (Participants) | 21
units on a scale | 16.14 (9.84)

3. Secondary Outcome: Change in Patient-rated Depression Severity
Description: Change in depression severity measured by the patient-rated Quick Inventory of Depressive Symptoms, Self-Rated (QIDS-SR16). The QIDS-SR16 is a self-report measure of depression severity with a range of 0-27, with higher scores indicative of more severe depression.
Time Frame: Assessed every 2 weeks from baseline to week 12, change from baseline to week 12 is reported
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Sertraline
Number analyzed (Participants) | 17
units on a scale | 3.82 (6.04)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Adverse events and serious adverse event definitions are concordant with clinicaltrials.gov definitions.
  Adverse events were assessed at every contact by asking individuals about any medical problems or potential side effects they were experiencing.
Arm/Group | Sertraline
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 14/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sertraline (N=21)
Upper Respiratory Infection (Infections and infestations) | 2
Vision changes (Eye disorders) | 1
Dry Eyes (Eye disorders) | 1
Vivid Dreams (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 1
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dry Mouth (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 3
Sexual Dysfunction (Reproductive system and breast disorders) | 2

LIMITATIONS AND CAVEATS:
Limitations include a small sample that reflects this is a pharmacoimaging study using MRI to examine imaging findings related to antidepressant treatment outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No